CLINICAL TRIAL: NCT02652637
Title: MOBILE Trial. Mechanical and Oral Antibiotic Bowel Preparation Versus no Bowel preparatIon for eLEctive Colectomy - a Multicenter, Prospective, Randomized, Controlled Trial.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Ville Sallinen, MD, PhD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HYKS-MOBILE
Record Dates: First submitted 2016-01-08; First posted 2016-01-12 (Estimated); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Colorectal Surgery
MeSH Terms: interventions — Neomycin; Metronidazole; Polyethylene Glycols

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Mechanical and oral antibiotic bowel preparation (Experimental): Mechanical bowel preparation using PEG, neomycin 2g p.o. (single-dose), and metronidazole 2g p.o. (single dose) are given the day before surgery.
  Interventions: Drug: neomycin, metronidazole, polyethylene glycol (PEG)
- No bowel preparation (No Intervention): No mechanical bowel preparation or oral antibiotics.

INTERVENTIONS:
Drug: neomycin, metronidazole, polyethylene glycol (PEG)
  Arms: Mechanical and oral antibiotic bowel preparation

SUMMARY:
Enchanced recovery after surgery (ERAS) protocols aim to provide safer and quicker recovery postoperatively. One of the elements in ERAS protocols is that bowel is not prepared before colorectal surgery. However, several recent retrospective register studies have suggested that mechanical bowel preparation combined to oral antibiotics before colectomy reduces complications compared to no preparation at all. This trial compares these two strategies to find out whether complications can indeed be reduced by mechanically preparing the bowel with oral antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing colon resection

Exclusion Criteria:

* Emergency surgery needed
* Bowel obstruction
* Colonoscopy scheduled to be undertaken peroperatively
* Other reason indicating mechanical preparation or contradicting it
* Allergy to used drugs (PEG, neomycin, metronidazole)

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Surgical site infection (CDC criteria) | 30 days from operation

SECONDARY OUTCOMES:
Comprehensive Complication Index | 30 days from operation
Anastomotic dehiscence | 30 days from operation
Reoperations | 30 days from operation
Readmissions | 30 days from operation
Length of hospital stay | During hospital stay, anticipated 2-30 days
Mortality | 30- and 90-days from operation
Adverse effects of antibiotics (diarrhea, clostridium) | 30 days from operation
Patients receiving adjuvant therapy divided by patients needing adjuvant therapy | 6 months from operation

OTHER OUTCOMES:
5-year overall survival | 5 years from operation
5-year disease specific survival | 5 years from operation
5-year recurrence free survival | 5 years from operation

CONTACTS AND LOCATIONS:
Locations (4):
- Finland (4):
  - Helsinki University Central Hospital, Helsinki
  - Central Finland Central Hospital, Jyväskylä
  - Oulu University Hospital, Oulu
  - Seinäjoki Central Hospital, Seinäjoki

REFERENCES:
- [Derived] Koskenvuo L, Lehtonen T, Koskensalo S, Rasilainen S, Klintrup K, Ehrlich A, Pinta T, Scheinin T, Sallinen V. Mechanical and oral antibiotic bowel preparation versus no bowel preparation for elective colectomy (MOBILE): a multicentre, randomised, parallel, single-blinded trial. Lancet. 2019 Sep 7;394(10201):840-848. doi: 10.1016/S0140-6736(19)31269-3. Epub 2019 Aug 8. PMID 31402112